CLINICAL TRIAL: NCT02131376
Title: Investigating a Novel Modifiable Factor Affecting Renal Function After Partial Nephrectomy: Cortical Renorrhaphy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual, interim analysis showed no statistical significance
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Chandru Sundaram, Professor of Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IUCRO-0459
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Renal Cell Carcinoma
Keywords: carcinoma, renal cell; partial nephrectomy; kidney function test; robotics
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cortical renorrhaphy (Active Comparator): Cortical renorrhaphy is performed after partial nephrectomy using a running barbed suture on MH (36mm) needle. Polymer locking clips are used to maintain tension. A base layer running stitch is performed prior to the cortical renorrhaphy.
  Interventions: Procedure: Renorrhaphy
- Non-renorrhaphy (Experimental): The suture closure of the renal cortex after tumor removal is omitted. A base layer running stitch only is performed for hemostasis and urine leak prevention.
  Interventions: Procedure: Non-renorrhaphy

INTERVENTIONS:
Procedure: Non-renorrhaphy — The suture closure of the renal cortex after tumor removal is omitted. A base layer running stitch only is performed for hemostasis and urine leak prevention.
  Other Names: renal reconstruction
  Arms: Non-renorrhaphy
Procedure: Renorrhaphy — After tumor resection the patient will have both a deep and cortical layer reconstruction
  Other Names: renal reconstruction
  Arms: Cortical renorrhaphy

SUMMARY:
Preserving kidney function during removal of a kidney tumor is becoming increasingly important as rates of chronic kidney disease increase. A novel modifiable factor (suture closure of the defect caused by tumor removal) was discovered on retrospective studies to account for nearly two-thirds of the 15% volume loss commonly seen in operated kidneys. We hypothesize that a randomized controlled surgical trial will show that omitting the suture closure both preserves renal function and will not lead to unreasonable postoperative complications.

DETAILED DESCRIPTION:
Purpose: To evaluate a never before studied modifiable factor affecting renal function after partial nephrectomy: the suture closure of the renal cortex after tumor removal (renorrhaphy).

Background:

There is increasing interest in preserving renal function when removing renal tumors. This is partly due to studies that link chronic kidney disease with cardiovascular events and overall survival. There is an approximate loss of 10% overall renal function after partial nephrectomy along with a loss of 15% of the volume in the operated kidney. Studies point to 3 factors leading to this loss in renal function after partial nephrectomy: 1) Poor preoperative renal function, 2) Ischemia time (clamping the renal blood vessels to decrease bleeding during surgery, and 3) Loss in renal volume from the surgery.

The only factor that is considered modifiable is ischemia time, especially when over 20-25-minutes in duration. Modern techniques now aid in keeping the ischemia time below the 25-minute cutoff. Leading experts from institutions such as the Cleveland Clinic, The University of Southern California, and The Mayo Clinic have concluded that the most important factor in preserving renal function, renal volume loss, is not modifiable.

Specific Aims: Our question is: if we are removing non-functional tissue (tumor) then why is there a loss in renal volume (15%) and function (10%)? We hypothesize that by omitting one particular step during surgery, sewing closed the defect caused by tumor removal, we will be able to improve renal volume loss and function (RENORRHAPHY CLIP http://youtu.be/NXOtUHdigj4). Indiana University is in a unique position to study this hypothesis as two of our surgeons have routinely omitted closing the defect left after tumor removal (NO RENORRHAPHY CLIP http://youtu.be/ZisMjrm85s8).

In a recently accepted abstract, we discovered that omitting the cortical closure (n=28) resulted in a 0.8% loss in glomerular filtration rate while using the closure resulted in a 7.3% loss (p=0.03). Following this discovery a 3D modeling project was performed to isolate the volume loss in operated kidneys using pre- and postoperative CT scans (not yet published). In this study, we discovered a 15% volume loss with cortical closure (n=38) compared to only a 5% loss without closure (n=20, p < 0.001).

Bias and confounders cannot completely be removed from our retrospective data making it hard to believe that others will consider our hypothesis without a randomized controlled trial (RCT). We propose a RCT for robotic partial nephrectomy (20 stitch closure vs. 20 no stitch closure) with the primary outcome being volume change in the affected kidney.

ELIGIBILITY:
3.0 INCLUSION/EXCLUSION CRITERIA

3.1 Inclusion criteria:

* ≥ 18 years of age.
* Must provide written informed consent
* Presence of cT1 renal mass by diagnostic CT assessment.
* Scheduled for partial nephrectomy of renal mass.
* Expected survival of at least 3 months.
* ECOG ≤ 1.
* Negative serum/urine pregnancy test within 24 hours for females of child bearing age prior to surgery
* Recovered from toxicity of any prior therapy to grade 1 or better
* If biopsy of mass has been done, pathology must be consistent with RCC.

3.2 Exclusion criteria:

* Solitary kidney
* Multiple or bilateral renal masses when more than one mass is operated on at the same time or within 4-months of each other.
* Hepatic or renal toxicity (GFR <30) greater than or equal to Grade 2 (using CTCAE version 4 standard definitions)
* Bleeding diathesis or inability to hold anticoagulation for surgery
* Participation in another investigational trial concurrently or within 30 days
* Significant acute or chronic medical, neurologic, or psychiatric illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
%Loss renal volume | 4months
  % loss in renal volume (cm3) of the operated kidney (post-operative CT at 4 mo vs. - pre-operative CT) using Phillips IntelliSpace portal semi-automated segmentation algorithm.

SECONDARY OUTCOMES:
Operative and postoperative complications | through 4months
  Operative and postoperative complications (urine leak, bleeds) through the 4month follow-up
Resistive index | In the operating room prior to resection (baseline) and immediately after resection of tumor
  This is a "change" outcome measure. Pre and post-partial nephrectomy on the day of surgery Doppler/US arterial resistive index changes are recorded.
Surgeon survey | immediately after surgery is complete
  Postoperative surgeon survey evaluating comfort with surgery-Likert scale questionnaire
Predicted volume loss | 4months
  Assess the volume loss predicted by a preoperative scoring system. The preoperative volume loss prediction will be compared to the 4month volume loss calculation based on CT scans.
%Loss in GFR | 4months
  % eGFR loss from pre to postoperative (4mo) followup
Adverse events as defined by the Clavien-Dindo classification system. | Through 4months

CONTACTS AND LOCATIONS:
Overall Officials: Chandru P Sundaram, MD, Principal Investigator — Indiana University Health; Clinton D Bahler, MD, Principal Investigator — Indiana University Health
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States